CLINICAL TRIAL: NCT00718003
Title: Noninvasive Examination of the Work of Breathing in Patients With Amyotrophic Lateral Sclerosis (ALS).
Status: Terminated | Type: Observational
Why Stopped: Terminated due to difficulty enrolling subjects.
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-15860
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.

SUMMARY:
The literature to date indicates that noninvasive positive pressure ventilation (NIPPV) provides effective noninvasive ventilator support, prolongs survival, and improves quality of life (QOL) in Amyotrophic Lateral Sclerosis (ALS) patients. It is generally recommended to patients when their pulmonary function testing demonstrates a drop to 50% forced vital capacity (FVC). One result of using NIPPV may be a reduction in the work of the breathing which would lead to decreased caloric needs. However, the work of breathing and the effects of noninvasive ventilation on caloric use have not been studied in patients with ALS. This is extremely important since there may be a reduction in the caloric needs when ALS patients are placed on NIPPV and if the caloric intake is not adjusted, overfeeding can occur. Overfeeding with too many calories can lead to an increase in carbon dioxide which would actually worsen the respiratory failure.

The overall aim of this project is to evaluate how many calories are used by ALS patients while at rest, when placed on NIPPV, and when breathing against a resistance. This will be accomplished using a metabolic cart during these activities. At present, the metabolic cart is routinely used in ALS patients at the time of feeding tube placement to calculate caloric needs. Using the cart to calculate the caloric expenditure on and off the ventilator will aid in calculating the work of breathing and the effects of NIPPV on work of breathing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with probable or definite ALS by El Escorial Criteria between ages 20-85 will be included for evaluation. They must have progression of disease over the preceding 6 months and duration of disease less then 5 years.

Exclusion Criteria:

* Patients who do not meet clinical criteria of the diagnosis including those with pure upper motor neuron syndromes (PLS) or pure lower motor syndromes (SMA, Multifocal conduction block, motor neuropathies).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Calories Used with and without NIPPV | 20 minutes
  Indirect calorimetry will be performed using a metabolic cart to determine caloric use over a 20 minute period without NIPPV. Following this, the test will be repeated over a 20 minute period with NIPPV.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Heiman-Patterson, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States